CLINICAL TRIAL: NCT05752136
Title: Preoperative Short-course Radiation Followed by Envafolimab Plus CAPEOX for MSS Locally Advanced Rectal Adenocarcinoma: a Prospective, Multicenter, Randomized Controlled Study (PRECAM-R)
Brief Title: Preoperative Short-course Radiation Followed by Envafolimab Plus CAPEOX for MSS Locally Advanced Rectal Adenocarcinoma
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sir Run Run Shaw Hospital (Other)
Responsible Party: Principal Investigator, Sheng Dai, Principal Investigator, head of medical affairs, Sir Run Run Shaw Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LXSHYJ-20221129-02
Record Dates: First submitted 2023-02-20; First posted 2023-03-02 (Actual); Last update posted 2023-05-08 (Actual); Status verified 2023-05

CONDITIONS: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms | interventions — envafolimab

STUDY DESIGN:
Intervention Model Description: The 54 enrolled patients with MSS-type advanced middle-low rectal cancer will receive a combined regimen of neoadjuvant chemoradiotherapy combined with immunotherapy and total mesorectal excision (TME surgery).
  The other 54 patients with MSS-type advanced middle-low rectal cancer will receive a combined regimen of neoadjuvant chemoradiotherapy combined with immunotherapy and total mesorectal excision (TME surgery).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neoadjuvant chemoradiotherapy combined with immunotherapy and total mesorectal excision (Experimental): Drug: Envafolimab This product is administered by subcutaneous injection. The recommended dose of subcutaneous injection is 150 mg, administered weekly (QW).
  Other Name: KN053
  Drug: Oxaliplatin 130mg/m2，ivgtt，d1
  Drug: Capecitabine 1000mg/m2，po，bid，d1-14
  Radiation: Short-course Radiation Short-course radiotherapy, using three-dimensional conformal or intensity-modulated radiotherapy, the dose is divided into 5Gy/f, the total dose is 25Gy/5f, 1f/d, and the irradiation is completed within 7 days.
  Procedure: TME surgery, total mesorectal excision The surgical method can choose open, laparoscopic or robotic according to the specific condition of the patient.
  Interventions: Biological: Envafolimab
- Neoadjuvant chemoradiotherapy and total mesorectal excision (No Intervention): Drug: Oxaliplatin 130mg/m2，ivgtt，d1
  Drug: Capecitabine 1000mg/m2，po，bid，d1-14
  Radiation: Short-course Radiation Short-course radiotherapy, using three-dimensional conformal or intensity-modulated radiotherapy, the dose is divided into 5Gy/f, the total dose is 25Gy/5f, 1f/d, and the irradiation is completed within 7 days.
  Procedure: TME surgery, total mesorectal excision The surgical method can choose open, laparoscopic or robotic according to the specific condition of the patient.

INTERVENTIONS:
Biological: Envafolimab — This product is administered by subcutaneous injection. The recommended dose of subcutaneous injection is 150 mg, administered weekly (QW).
  Arms: Neoadjuvant chemoradiotherapy combined with immunotherapy and total mesorectal excision

SUMMARY:
Short-course radiotherapy combined with immunotherapy may bring revolutionary changes to the preoperative neoadjuvant treatment mode for locally advanced rectal cancer.In view of the shortcomings of the current preoperative neoadjuvant treatment model for locally advanced rectal cancer, we will explore the feasibility of a new model of short-course radiotherapy combined with immunotherapy, and develop a possible optimal plan based on the existing theoretical basis, namely "short-course radiotherapy + PD-L1 monoclonal antibody combined with CAPEOX chemotherapy for 2 cycles", and explore the efficacy and adverse effects of this model. The study will also attempt to explore the characteristics of the treatment beneficiary population, explore the characteristics of the treatment beneficiary population by multi-dimensional tumor and microenvironmental information through multi-omics sequencing analysis, attempt to build an efficacy prediction model, early screening of the treatment beneficiary population for precise treatment, and thus explore a new model of radiotherapy combined with immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are willing to receive neoadjuvant therapy.
2. ≧18 years old.
3. Diagnosed by digital rectal examination, colonoscopy, and high-resolution MRI of the pelvis, the tumor is less than or equal to 12 cm from the anus.
4. Histologically diagnosed as rectal adenocarcinoma.
5. The clinical staging by pelvic contrast-enhanced CT and pelvic high-resolution MRI were cT2-4a N+, cT3/T4a N0.
6. MMR protein detection or MSI gene detection of rectal cancer specimens confirmed pMMR or MSS before treatment .
7. The patient has good compliance and can come to the hospital for re-examination as required.
8. ECOG Scale of Performance Status score 0-1 point.
9. Have not received anti-tumor and immunotherapy before enrollment.
10. Laboratory inspections must meet the following standards:

    * White blood cell count>3.5×109/L, absolute value of neutrophils>1.8×109/L, platelet count ≥75×109/L, hemoglobin ≥100g/L;

      * INR≤1.5, and APTT≤1.5 times the upper limit of normal or partial prothrombin time (PT) ≤1.5 times the upper limit of normal;

        * Total bilirubin ≤ 1.25 times the upper limit of normal; ALT and AST < 5 times the upper limit of normal;

          * 24h creatinine clearance >50mL/min or serum creatinine <1.5 times the upper limit of normal.
11. Voluntarily participate in this study and sign the informed consent.

Exclusion Criteria:

1. History of other malignant diseases in the past 5 years.
2. Patients with metastases from other sites (stage IV patients).
3. Patients with clinical staging of T1-2N0 or T4b, or positive lateral lymph nodes by pelvic contrast-enhanced CT and pelvic high-resolution MRI.
4. Patients with intestinal obstruction, intestinal perforation, intestinal bleeding, etc. requiring emergency surgery.
5. Known allergic to oxaliplatin, capecitabine, PD-L1 monoclonal antibody and other drugs.
6. Pathologically suggested signet ring cell carcinoma and mucinous adenocarcinoma.
7. dMMR or MSI-H patients.
8. The patient is accompanied by any unstable systemic disease, including but not limited to: severe infection, uncontrolled diabetes, hypertension uncontrolled by medication, unstable angina, cerebrovascular accident or transient cerebral ischemia, myocardial Infarction, congestive heart failure, severe cardiac arrhythmia requiring medication, hepatic, renal or metabolic disease; disease affecting the patient's life.
9. The disease (such as mental illness, etc.) or condition (such as alcoholism or drug abuse, etc.) associated with the patient will increase the risk of the patient receiving the trial drug treatment or affect the patient's compliance with the trial requirements, or may confuse the research results.
10. Active autoimmune disease that may worsen while receiving immunostimulants.
11. Known history of positive HIV test or known acquired immunodeficiency syndrome.
12. Patients who are using immunosuppressive agents, except for the following conditions:

    * Intranasal, inhaled, topical steroids, or topical steroid injections (eg, intra-articular injections);

      * Physiological doses of systemic corticosteroids ≤10 mg/day prednisone or equivalent;

        * Steroids used to prevent allergic reactions (eg, before CT scan).
13. Received any other experimental drug treatment or participated in another interventional clinical trial within 30 days before screening
14. Women who are pregnant or breastfeeding or who plan to become pregnant or breastfeeding during the study period; men or women who are unwilling to take effective contraceptive measures.
15. Vulnerable groups, including mentally ill, cognitively impaired, critically ill patients, minors, etc.
16. Other conditions that the investigator judges that the patient is not suitable to participate in the clinical study, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
pCR rate | Up to 10 weeks (once surgery is done) ]
  The primary objective of the study is to evaluate the pathologic complete response (pCR) rate following short-course radiation then Envafolimab Plus CAPEOX

SECONDARY OUTCOMES:
Tumor regression grade | Up to 10 weeks (once surgery is done)
  Tumor regression grade following short-course radiation then Envafolimab Plus CAPEOX as assessed by AJCC/CAP TRG system
OS | Up to 3 years
  The proportion of participants who remain survival at 3 years
PFS | Up to 3 years
  The proportion of participants who remain progression free at 3 years
TRAEs | Up to 3 years
  Number of participants with treatment-related adverse events as assessed by NCI-CTCAE v5.0
Surgical Complications | Up to 24 weeks
  Surgical Complications of total mesorectal resection procedure for patients after short-course radiation then Envafolimab Plus CAPEOX as assessed by Clavien-Dindo classification
QoL | Up to 3 years
  Quality of life of the patients in two neoadjuvant settings of short-course radiation followed with or without Envafolimab Plus CAPEOX as assessed by Functional Assessment of Cancer Therapy - Colorectal (FACT-C) questionnaire liscenced from The Functional Assessment of Chronic Illness Therapy System ("FACIT System"). By using the Manual scoring template, some items are reverse scored. Subscale scores, total scores and TOI scores. The higher the score, the better the QOL.

CONTACTS AND LOCATIONS:
Overall Officials: sheng dai, Principal Investigator — Sir Run Run Shaw Hospital
Locations (1):
- Sir Run Run Shaw Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided